CLINICAL TRIAL: NCT05091294
Title: Does the Injection Rate of Local Anesthetic Affect the Onset of Sensory Block and Incidence of Hypotension in Caesarean Section
Brief Title: The Effect of Injection Rate of Local Anesthetic in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ersagun Tugcugil, Ass. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-52; Ahmet Beşir (Other: KaradenizTU)
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia, Spinal; Anesthesia, Obstetrical
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S:33 (Active Comparator): 120-second local anesthesic (% 0,5 Bupivacaine) injection time
  Interventions: Other: Local anesthetic injection rate in spinal anesthesia
- Group F:34 (Active Comparator): 15-second local anesthesic(% 0,5 Bupivacaine) injection time
  Interventions: Other: Local anesthetic injection rate in spinal anesthesia

INTERVENTIONS:
Other: Local anesthetic injection rate in spinal anesthesia — Administering intrathecal local anesthetics for all patients according to height and weight.

SUMMARY:
This randomized double-blind study aimed to compare the effects of two different subaracnoid lokal anesthetic injection rate in cesarean section. Totally 67 patients were included. The groups were compared in terms of maximum sensory and motor block level, time to reach T6 level, hemodynamic changes and nausea- vomiting saved.

DETAILED DESCRIPTION:
A total of 67 patients 18-40 years undergoing cesarean, who were graded as American Society of Anesthesiologists physical status were randomly allocated into two groups, 120-sn injection time (n=34, Group F), 15-sn injection time (n=33, Group S). When the level of the sensory block achieve the T6 level the surgery was let to begin. The groups were compared in terms of hemodynamic values, use of efedrin, the time to achieve sensory block to the T6 level, maximum sensory block level and motor block level.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists risk score (ASA) I-II risk status
* Singleton pregnancy aged
* Between 18-40 years

Exclusion Criteria:

* Pregnant women with contraindications for spinal anesthesia;
* Placental anomaly;
* Hypertension
* Cardiac disease
* Vascular disease
* Hepatic disease
* Renal disease
* Hemodynamic instability
* Spinal deformity;
* Severe mental retardation
* Weight < 50 kg or >110 kg; height < 140 cm or > 180 cm
* Metabolic and Acid-base balance disorders
* Emergency patients

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All patients are pregnant.
Enrollment: 67 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
sensory block | 2 minutes interval
  The time to reach the sufficient sensory block and maximum level of sensory block was significantly shorter in Group S
Hypotension | 2 minutes interval
  The time to onset of hypotension was significantly shorter in Group F

CONTACTS AND LOCATIONS:
Overall Officials: Ersagun tugcugil, Principal Investigator — KARADENİZ TEKNİK ÜNİVERSİTESİ DEPARTMENT OF ANESTHESİOLOGİA AND REANİMATİON
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No